CLINICAL TRIAL: NCT02490891
Title: Study of the Angiogenesis Measured by PET/CT With 18F-RGD-K5 in Patients With Lymphoma : a Preliminary Study
Brief Title: Study of the Angiogenesis by PET/CT in Patients With Lymphoma
Acronym: RGDLymphome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Other
Other Study IDs: CHB14.02
Record Dates: First submitted 2015-07-01; First posted 2015-07-07 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma
Keywords: Lymphoma, angiogenesis, PET scan
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET scan with RGD K5 imaging (Experimental): PET scan with RGD K5 tracer will be performed before and after two cycles of chemotherapy
  Interventions: Device: RGD K5 PET scan

INTERVENTIONS:
Device: RGD K5 PET scan — PET scan with a tracer specific for angiogenesis (RGD K5) will be performed before and after 2 cycles of chemotherapy

SUMMARY:
The aim of the study is to measure tumoral angiogenesis modifications by RGD-K5 PET/CT before and after 2 cycles of chemotherapy in patients with lymphoma and a large tumoral mass

DETAILED DESCRIPTION:
After inclusion PET scans with FDG tracer and with a specific tracer of angiogenesis will be performed on patient with lymphoma. After two cycles of chemotherapy PET scans with the same tracers will be performed.

Overall survival and disease free survival will be monitored during 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age ≥ 18 years old
* OMS ≤ 1
* Histological diagnosis of diffuse large B-cell lymphoma what ever the subtype
* Presence of measurable tumor with at least a node mass superior to 3 centimeters
* Stage I to IV
* Inform consent signed

Exclusion Criteria:

* Primary cerebral lymphoma
* Absence of fixing on FDG-PET exam
* Pregnant , child bearing, breast feeding or without effective contraception method woman
* Hypersensitivity to RGD-K5
* Hypersensitivity to FDG
* Poorly controlled diabètes (glycemia ≥ 10 millimoles/liter)
* Neoplastic disease (less than 2 years or in progression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Measure of angiogenesis with RGD K5 PET scan | 3 months
  Measure of fixation, metabolic volume and angiogenic volume with RGD K5 traver

SECONDARY OUTCOMES:
Measure of angiogenic volume with K5 tracer | 3 months
  Measure of SUV max, SUV peak, SUV mean, metabolic volume and angiogenic volume to determine angiogenesis parameters with RGD-K5 PET scansand correlation with results of anatomopathology.
Overall survival | 18 months
  Time between inclusion and death whatever the cause
Disease-free survival | 18 months
  Time between inclusion and progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Vera, MD, PhD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France